CLINICAL TRIAL: NCT04527627
Title: Development and Evaluation of a Nursing Intervention in the Patient Being Discharged From the Intensive Care Unit: a Protocol for Mixed Methods Research
Brief Title: Nursing Intervention in the Patient Being Discharged From the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2016/0484
Record Dates: First submitted 2020-08-17; First posted 2020-08-26 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-08

CONDITIONS: Anxiety; Depression
Keywords: empowerment patient; patient education; icu discharge; nursing interventions; anxiety; depression; post-traumatic stress disorder; post icu syndrome
MeSH Terms: conditions — Anxiety Disorders; Depression; Patient Participation; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The nursing empowerment intervention will be administered in the experimental group
  Interventions: Behavioral: Nursing Empowerment Intervention
- Control Group (CG) (No Intervention): The nursing empowerment intervention will not be administered in the control group

INTERVENTIONS:
Behavioral: Nursing Empowerment Intervention — Nursing empowerment intervention The intervention will be carried out during the ICU discharge planning. A "Patient Information Guide for Intensive Care Unit patients" will be developed.
  The guide will be based on the findings obtained in a previous qualitative study and on previous studies on patient empowerment and education. Its structure will take into account the dimensions of empowerment: bio-physiological, functional, social, experience, ethics and the financial aspect. The guide will be reviewed by experts in the development of information guides for patients and family members and will be evaluated by the participating ICUs before use.
  EG patients will receive the intervention verbally and in booklet format from the study nurses at each ICU.
  Arms: Experimental Group (EG)

SUMMARY:
Background: Psychiatric disorders, such as anxiety, depression or post-traumatic stress disorder (PTSD), are common among critical disease survivors. Interventions aimed to decrease ICU impact on patient mental well-being are needed.

Methods/Design: The study will evaluate an educational nursing intervention addressed to ease the transition during ICU discharge by empowering the patient. A quantitative design will be used to measure the effectiveness of the nursing intervention through an experimental pre-test/post-test with control group design.

Participants will consist of patients from three critical care units from three different hospitals.

Data will be obtained from Hospital Anxiety and Depression Scale (HADS). Data will be analysed through descriptive and inferential statistics.

Discussion: This study will help to develop and implement an intervention to help patients lessen anxiety and depression associated to their transition from ICU to the general ward.

DETAILED DESCRIPTION:
Method An experimental pre-test-post-test design will be used. Setting and participants The study will be carried out in the ICU of three university hospitals which have 151 level 3 ICU beds and where the nurse/patient ratio is 1:2. The three ICUs admit approximately 2000 patients per year. Participants who meet the following inclusion criteria will be included: age > 18 years; ICU stay > 48h; speaker of one of the two official languages of the region and carrying out a personal interview, Glasgow Coma Score of 15, Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) negative, and provision of signed informed consent. Patients with a pre-admission diagnosis of mental illness will be excluded.

Patients will be selected by simple random probabilistic sampling. Patients will be recruited through the ICU admission list and randomly assigned to the experimental group (EG) and the control group (CG). To calculate the sample number needed, on the basis of a statistical power of 80% and a level of confidence of 95% in a unilateral analysis, and estimating the percentage of patients who have high anxiety at ICU discharge at 50% (between 30% and 75% according to reports), a sample of 86 patients per group will be needed (assuming 15% losses per group) to detect a difference of >20% as statistically significant (expected to be 0.5 for the CG and 0.28 for the EG).

Nursing empowerment intervention The intervention will be carried out during the ICU discharge planning. A "Patient Information Guide for Intensive Care Unit patients" will be developed.

The guide will be based on the findings obtained in a previous qualitative study and on previous studies on patient empowerment and education. The guide structure will take into account the dimensions of empowerment: bio-physiological, functional, social, experience, ethics and the financial aspect. The guide will be reviewed by experts in the development of information guides for patients and family members and will be evaluated by the participating ICUs before use.

EG patients will receive the intervention verbally and in booklet format from the study nurses at each ICU. CG patients will receive the usual nursing treatment provided during ICU discharge, which usually consists of verbal information about the time and place of destination.

Variables:

1. Independent variable: Nursing empowerment intervention administered to the patient during ICU discharge.
2. Dependent variable: Level of anxiety and depression (HADS scale) pre-post ICU discharge.
3. Sociodemographic variables: sex (male/female), age (in years), educational level (none, primary, secondary, higher), profession, family situation (lives alone, with family or friends) and marital status (single, married or cohabiting, widower, divorced).
4. Clinical variables: severity level (APACHE II), reason for ICU admission and days of stay in the ICU.

Data will be collected using a first contact with the patient in the ICU, and the study objectives and informed consent will be explained.

The researcher will administer the HADS scale to the EG and CG groups before ICU discharge and after ICU discharge (in the destination ward).

Instruments:

1. Glasgow Coma Score: The Glasgow scale is designed to assess the level of consciousness, and includes the assessment of the ocular, verbal and motor response. It is simple, objective and easily reproducible.
2. The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) adapted and translated to Spanish by Tobar et al. (2010), which is recommended and validated in the detection of delirium. The four criteria that characterize delirium are evaluated using four questions for each area (change in mental status, inattention, altered consciousness and disorganized thinking).
3. Hospital Anxiety and Depression Scale (HADS): Adapted and validated in Spanish by Tejero, Guimera, Farré and Peri (1986) it comprises two subscales of 7 items each, one for anxiety and one for depression. The intensity/frequency of symptoms is evaluated on a four-point Likert scale. For each subscale, the score ranges from 0 to 21, with the following cut-off points: 0-7 Normal; 8-10 Doubtful/possible clinical problem; >10 Likely clinical problem. The HADs measures the current status during the last week. Designed to be administered to subjects with organic diseases, the physical aspects that may accompany anxiety or depression have been eliminated, leaving the emotional aspects ones. In addition to the quantitative evaluation, it may be stratified into non-anxious or non-depressed if the HADS scores are < 8; possible or doubtful between 8 and 10, and likely or affirmative if they are ≥ 11. The authors consider that, for research purposes, if a low proportion of false positives are to be obtained, the upper limit with values of 10 or 11 should be used, while values of 8 or 9 would prevent false negatives. For this study, a value of 10 was decided on as a cut-off point between the presence or absence of anxiety and depression.
4. Acute Physiology and Chronic Health Evaluation (APACHE) II: To measure and evaluate the severity of the critically ill, Knaus produced in 1981 the first version, comprising 34 items, which were reduced reducing to 14 in the second version in 1985. APACHE II classifies disease severity using 12 usual physiological measures, the previous health status and age, with a score ranging from 0 to 71 points.

Data analysis The data will be analysed using the SPSS v23 statistical package. A descriptive analysis of the study variables will be made (means and standard deviation and medians and 25-75 percentiles (IQR) for quantitative variables according to the normality of distribution, and frequencies and percentages for qualitative variables). The possible relationship between sociodemographic and clinical variables and the level of anxiety and depression will be analysed using Pearson's correlation coefficient, the Student's t test and ANOVA or their nonparametric equivalents based on the type of variable and its distribution and the number of subgroups compared. The chi square test will be used to compare the variation in categorical variables between the EG and CG. The Mann-Whitney test or the Wilcoxon test will be used to compare the mean anxiety scale score between EG and CG. Statistical significance will be established as p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ICU stay > 48h
* Speaker of one of the two official languages of the region Catalan or Spanish and carrying out a personal interview
* Glasgow Coma Score of 15
* Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) negative
* Provision of signed informed consent

Exclusion Criteria:

- Pre ICU admission diagnosis of mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Level of anxiety and depression assessed by Hospital Anxiety and Depression Scale. | 1 week
  The outcome 1 will be mesured with the anxiety and depression scale (HADS) after ICU discharge. The HADS measures the current status during the last week. A value of 10 is the cut-off point between the presence or absence of anxiety and depression.

SECONDARY OUTCOMES:
Level of anxiety and depression at ICU discharge assessed by Hospital Anxiety and Depression Scale | Up to 2 days
  The outcome 2 will be mesured with the anxiety and depression scale (HADS) during ICU discharge. The HADS measures the current status during the last week. A value of 10 is the cut-off point between the presence or absence of anxiety and depression.
Level of anxiety and depression at the general ward stay assessed by Hospital Anxiety and Depression Scale | After 2 days
  The outcome 3 will be mesured with the anxiety and depression scale (HADS) at the general ward. The HADS measures the current status during the last week. A value of 10 is the cut-off point between the presence or absence of anxiety and depression.
Severity level at ICU admission assessed by Acute Physiology and Chronic Health Evaluation (APACHE) II | Day 1
  APACHE II is a clinical variable. It will be used to measure and evaluate the severity of the critically ill. It classifies disease severity using 12 usual physiological measures, the previous health status and age, with a score ranging from 0 to 71 points.
Duration of ICU stay | Up to 60 days
  Duration of ICU stay is a clinical variable. This variable indicates how many days the patients needs to recovery from critically ill.
Sex: male or female | Day 1
  Sex is a sociodemographic variable. Acording to the literature, female sex presents more ansiety and depression than male sex.
Age in years | Day 1
  Sociodemographic variable
Educational level: none, primary, secondary or higher | Day 1
  Sociodemographic variable
Family situation: lives alone, with family or friends | Day 1
  Sociodemographic variable
Marital status: single, married, cohabiting, widower or divorced | Day 1
  Sociodemographic variable

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Cuzco, RN, Principal Investigator — Hospital Clínic of Barcelona; Pedro Castro, MD, Study Director — Hospital Clínic of Barcelona; Pilar Delgado-Hito, RN, Study Director — University of Barcelona
Locations (3):
- Spain (3):
  - Hospital de Bellvitge, Barcelona, Hospitalet de Llobregat
  - Hospital Clínic of Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Result] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Result] Svenningsen H, Langhorn L, Agard AS, Dreyer P. Post-ICU symptoms, consequences, and follow-up: an integrative review. Nurs Crit Care. 2017 Jul;22(4):212-220. doi: 10.1111/nicc.12165. Epub 2015 Feb 17. PMID 25688675
- [Result] Fumis RR, Ranzani OT, Martins PS, Schettino G. Emotional disorders in pairs of patients and their family members during and after ICU stay. PLoS One. 2015 Jan 23;10(1):e0115332. doi: 10.1371/journal.pone.0115332. eCollection 2015. PMID 25616059
- [Result] Milton A, Bruck E, Schandl A, Bottai M, Sackey P. Early psychological screening of intensive care unit survivors: a prospective cohort study. Crit Care. 2017 Nov 9;21(1):273. doi: 10.1186/s13054-017-1813-z. PMID 29121983
- [Result] Ferrand N, Zaouter C, Chastel B, Faye K, Fleureau C, Roze H, Dewitte A, Ouattara A. Health related quality of life and predictive factors six months after intensive care unit discharge. Anaesth Crit Care Pain Med. 2019 Apr;38(2):137-141. doi: 10.1016/j.accpm.2018.05.007. Epub 2018 Jun 1. PMID 29864552
- [Result] Thomas S, Mehrholz J. Health-related quality of life, participation, and physical and cognitive function of patients with intensive care unit-acquired muscle weakness 1 year after rehabilitation in Germany: the GymNAST cohort study. BMJ Open. 2018 Jul 13;8(7):e020163. doi: 10.1136/bmjopen-2017-020163. PMID 30007926
- [Result] de Grood C, Leigh JP, Bagshaw SM, Dodek PM, Fowler RA, Forster AJ, Boyd JM, Stelfox HT. Patient, family and provider experiences with transfers from intensive care unit to hospital ward: a multicentre qualitative study. CMAJ. 2018 Jun 4;190(22):E669-E676. doi: 10.1503/cmaj.170588. PMID 29866892
- [Result] Stelfox HT, Lane D, Boyd JM, Taylor S, Perrier L, Straus S, Zygun D, Zuege DJ. A scoping review of patient discharge from intensive care: opportunities and tools to improve care. Chest. 2015 Feb;147(2):317-327. doi: 10.1378/chest.13-2965. PMID 25210942
- [Result] Won MH, Son YJ. Development and psychometric evaluation of the Relocation Stress Syndrome Scale-Short Form for patients transferred from adult intensive care units to general wards. Intensive Crit Care Nurs. 2020 Jun;58:102800. doi: 10.1016/j.iccn.2020.102800. Epub 2020 Jan 18. PMID 31964557
- [Result] Nikayin S, Rabiee A, Hashem MD, Huang M, Bienvenu OJ, Turnbull AE, Needham DM. Anxiety symptoms in survivors of critical illness: a systematic review and meta-analysis. Gen Hosp Psychiatry. 2016 Nov-Dec;43:23-29. doi: 10.1016/j.genhosppsych.2016.08.005. Epub 2016 Aug 28. PMID 27796253
- [Result] Hatch R, Young D, Barber V, Griffiths J, Harrison DA, Watkinson P. Anxiety, Depression and Post Traumatic Stress Disorder after critical illness: a UK-wide prospective cohort study. Crit Care. 2018 Nov 23;22(1):310. doi: 10.1186/s13054-018-2223-6. PMID 30466485
- [Derived] Cuzco C, Castro P, Marin Perez R, Ruiz Garcia S, Nunez Delgado AI, Romero Garcia M, Martinez Momblan MA, Benito Aracil L, Carmona Delgado I, Canalias Reverter M, Nicolas JM, Martinez Estalella G, Delgado-Hito P. Impact of a Nurse-Driven Patient Empowerment Intervention on the Reduction in Patients' Anxiety and Depression During ICU Discharge: A Randomized Clinical Trial. Crit Care Med. 2022 Dec 1;50(12):1757-1767. doi: 10.1097/CCM.0000000000005676. Epub 2022 Sep 30. PMID 36178294
- [Derived] Cuzco C, Castro Rebollo P, Marin Perez R, Nunez Delgado AI, Romero Garcia M, Martinez Momblan MA, Estrada Reventos D, Martinez Estalella G, Delgado-Hito P. Mixed-method research protocol: Development and evaluation of a nursing intervention in patients discharged from the intensive care unit. Nurs Open. 2021 Nov;8(6):3666-3676. doi: 10.1002/nop2.894. Epub 2021 May 6. PMID 33955196